CLINICAL TRIAL: NCT00642941
Title: A Phase II Trial of R1507, a Recombinant Human Monoclonal Antibody to the Insulin-Like Growth Factor-1 Receptor for the Treatment of Participants With Recurrent or Refractory Ewing's Sarcoma, Osteosarcoma, Synovial Sarcoma, Rhabdomyosarcoma and Other Sarcomas.
Brief Title: A Study of R1507 in Participants With Recurrent or Refractory Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed to further enrollment due to the decision by the Sponsor to discontinue development of R1507.
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Sarcoma Alliance for Research through Collaboration (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO21157; SARC011; 2007-003940-30 (EudraCT Number); NCT00615680 (obsolete NCT alias)
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — RG-1507 monoclonal antibody

ARMS (12):
- Cohort 1: Ewings Sarcoma Primary Cohort (Experimental): Participants 2 years of age and older with recurrent or refractory sarcoma receive R1507 as 9 mg/kg via IV infusion once weekly until disease progression, intercurrent illness, unacceptable toxicity, prolonged (2-week) time off treatment, withdrawal, loss to follow-up, investigator decision, or death. Cohort 1 includes individuals with Ewing's sarcoma who have relapsed within 24 weeks after diagnosis and have received two or more prior chemotherapy regimens.
  Interventions: Drug: RG1507
- Cohort 2: Ewings Sarcoma Secondary Cohort (Experimental): Participants 2 years of age and older with recurrent or refractory sarcoma receive R1507 as 9 mg/kg via IV infusion once weekly until disease progression, intercurrent illness, unacceptable toxicity, prolonged (2-week) time off treatment, withdrawal, loss to follow-up, investigator decision, or death. Cohort 2 includes individuals with Ewing's sarcoma who have relapsed more than 24 weeks after diagnosis and have only received one prior chemotherapy regimen.
  Interventions: Drug: RG1507
- Cohort 3: Ewings Sarcoma Expanded Cohort (Experimental): Participants 2 to 21 years of age with recurrent or refractory sarcoma receive R1507 as 27 mg/kg via IV infusion every 3 weeks until disease progression, intercurrent illness, unacceptable toxicity, prolonged (2-week) time off treatment, withdrawal, loss to follow-up, investigator decision, or death. Cohort 3 includes individuals with Ewing's sarcoma who were enrolled and treated following safety evaluation in other cohorts.
  Interventions: Drug: RG1507
- Cohort 4: Osteosarcoma (Experimental): Participants 2 years of age and older with recurrent or refractory sarcoma receive R1507 as 9 mg/kg via IV infusion once weekly until disease progression, intercurrent illness, unacceptable toxicity, prolonged (2-week) time off treatment, withdrawal, loss to follow-up, investigator decision, or death. Cohort 4 includes individuals with osteosarcoma.
  Interventions: Drug: RG1507
- Cohort 5: Synovial Sarcoma (Experimental): Participants 2 years of age and older with recurrent or refractory sarcoma receive R1507 as 9 mg/kg via IV infusion once weekly until disease progression, intercurrent illness, unacceptable toxicity, prolonged (2-week) time off treatment, withdrawal, loss to follow-up, investigator decision, or death. Cohort 5 includes individuals with synovial sarcoma.
  Interventions: Drug: RG1507
- Cohort 6: Rhabdomyosarcoma (Experimental): Participants 2 years of age and older with recurrent or refractory sarcoma receive R1507 as 9 mg/kg via IV infusion once weekly until disease progression, intercurrent illness, unacceptable toxicity, prolonged (2-week) time off treatment, withdrawal, loss to follow-up, investigator decision, or death. Cohort 6 includes individuals with rhabdomyosarcoma.
  Interventions: Drug: RG1507
- Cohort 7a: Alveolar Soft Part Sarcoma (Experimental): Participants 2 years of age and older with recurrent or refractory sarcoma receive R1507 as 9 mg/kg via IV infusion once weekly until disease progression, intercurrent illness, unacceptable toxicity, prolonged (2-week) time off treatment, withdrawal, loss to follow-up, investigator decision, or death. Cohort 7a includes individuals with alveolar soft part sarcoma.
  Interventions: Drug: RG1507
- Cohort 7b: Desmoplastic Small Round Cell Tumors. (Experimental): Participants 2 years of age and older with recurrent or refractory sarcoma receive R1507 as 9 mg/kg via IV infusion once weekly until disease progression, intercurrent illness, unacceptable toxicity, prolonged (2-week) time off treatment, withdrawal, loss to follow-up, investigator decision, or death. Cohort 7b includes individuals with desmoplastic small round cell tumors.
  Interventions: Drug: RG1507
- Cohort 7c: Extraskeletal Myxoid Chondrosarcoma (Experimental): Participants 2 years of age and older with recurrent or refractory sarcoma receive R1507 as 9 mg/kg via IV infusion once weekly until disease progression, intercurrent illness, unacceptable toxicity, prolonged (2-week) time off treatment, withdrawal, loss to follow-up, investigator decision, or death. Cohort 7c includes individuals with extraskeletal myxoid chondrosarcoma.
  Interventions: Drug: RG1507
- Cohort 7d: Clear Cell Sarcoma (Experimental): Participants 2 years of age and older with recurrent or refractory sarcoma receive R1507 as 9 mg/kg via IV infusion once weekly until disease progression, intercurrent illness, unacceptable toxicity, prolonged (2-week) time off treatment, withdrawal, loss to follow-up, investigator decision, or death. Cohort 7d includes individuals with clear cell sarcoma.
  Interventions: Drug: RG1507
- Cohort 7e: Myxoid Liposarcoma (Experimental): Participants 2 years of age and older with recurrent or refractory sarcoma receive R1507 as 9 mg/kg via IV infusion once weekly until disease progression, intercurrent illness, unacceptable toxicity, prolonged (2-week) time off treatment, withdrawal, loss to follow-up, investigator decision, or death. Cohort 7e includes individuals with myxoid liposarcoma.
  Interventions: Drug: RG1507
- Cohort 8: Diagnosis Not Specified (Experimental): Participants 2 years of age and older with recurrent or refractory sarcoma receive R1507 as 9 mg/kg via IV infusion once weekly until disease progression, intercurrent illness, unacceptable toxicity, prolonged (2-week) time off treatment, withdrawal, loss to follow-up, investigator decision, or death. Cohort 8 includes individuals with subtypes of sarcoma not specified in the protocol.
  Interventions: Drug: RG1507

INTERVENTIONS:
Drug: RG1507 — Participants will receive R1507 IV infusion as 9 mg/kg once weekly or 27 mg/kg every 3 weeks, depending upon the cohort in which the participants are enrolled.

SUMMARY:
The study was primarily designed to determine objective response, progression-free survival (PFS), and the safety and tolerability of R1507 in participants with recurrent or refractory Ewing's sarcoma, osteosarcoma, synovial sarcoma, rhabdomyosarcoma and other sarcomas including alveolar soft part sarcoma, desmoplastic small round cell tumor, extraskeletal myxoid chondrosarcoma, clear cell sarcoma, and myxoid liposarcoma.

ELIGIBILITY:
Inclusion Criteria:

* progressive, recurrent or refractory Ewing's sarcoma, or recurrent or refractory osteosarcoma, synovial sarcoma, rhabdomyosarcoma, or other sarcomas of the following sub-types: alveolar soft part sarcoma, desmoplastic small round cell tumor, extraskeletal myxoid chondrosarcoma, clear cell sarcoma and myxoid liposarcoma;
* Cohort 3 only: age must be >= 2 and <= 21 years

Exclusion Criteria:

* clinically significant unrelated systemic illness which would compromise the participant's ability to tolerate the investigational agent, or interfere with the study procedures or results;
* known hypersensitivity to any of the components of R1507 or prior hypersensitivity reactions to monoclonal antibodies;
* treatment (within the past 2 weeks) with pharmacologic doses of corticosteroids or other immunosuppressive agents;
* current or prior therapy with insulin-like growth factor (IGF) inhibitor (monoclonal or specific kinase inhibitor);
* history of solid organ transplant;
* other malignant disease diagnosed within the previous 5 years, excluding intra-epithelial cervical neoplasia or non-melanoma skin cancer;
* active central nervous system disease

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2007-12-18 (Actual); Primary Completion 2014-02-19 (Actual); Study Completion 2014-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (41):
- United States (22):
  - City of Hope National Medical Center, Duarte, California
  - UCLA School Of Medicine Mattel's Children's Hospital At UCLA; Division Of Hematology-Oncology, Los Angeles, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Stanford Comprehensive Cancer Center, Stanford, California
  - Washington Cancer Institute; Washington Hospital Center, Washington D.C., District of Columbia
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Johns Hopkins Hospital, Baltimore, Maryland
  - NIH/NCI, Bethesda, Maryland
  - Massachusetts General Hospital; Dana Farber Partnes Cancer Center, Boston, Massachusetts
  - Dana Farber Partners Can Ctr, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Nebraska Methodist Hospital; Onc Hem West, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Albert Einstein College of Medical Pediatrics; Department of Pediatrics, The Bronx, New York
  - Carolinas Hematology Oncology Associates; Investigational Drug Services - Pharmacy, Charlotte, North Carolina
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - Pennsylvania Oncology Hema Asc, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Texas Children's Cancer Center; Baylor College of Medicine, Houston, Texas
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute; Orthopedic Center, Salt Lake City, Utah
- Peter Maccallum Cancer Institute; Medical Oncology, Melbourne, Victoria, Australia
- BCCA-Vancouver Cancer Centre, Vancouver, British Columbia, Canada
- France (5):
  - Institut Bergonie; Oncologie, Bordeaux
  - Centre Oscar Lambret; Chir Cancerologie General, Lille
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Institut Curie; Oncologie Medicale, Paris
  - Institut Gustave Roussy; Service Pediatrique, Villejuif
- Germany (3):
  - HELIOS Klinikum Bad Saarow; Klinik für Innere Medizin III, Bad Saarow
  - Uniklinik Mannheim; Sektion Chirurgische Onkologie & Thoraxchirurgie, Mannheim
  - University Hospital Tübingen, Tübingen
- Italy (2):
  - Istituti Ortopedici Rizzoli, Bologna, Emilia-Romagna
  - Istituto Nazionale Tumori, Sarcoma Unit, Milan, Lombardy
- Erasmus Mc - Daniel Den Hoed Kliniek; Medical Oncology, Rotterdam, Netherlands
- Norwegian Radium Hospital, Oslo, Norway
- Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona, Spain
- Skånes University Hospital, Skånes Department of Onclology, Lund, Sweden
- United Kingdom (3):
  - UCL Hospital NHS Trust, London
  - Royal Marsden Hospital; Dept of Med-Onc, London
  - Christie Hospital NHS Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Asmane I, Watkin E, Alberti L, Duc A, Marec-Berard P, Ray-Coquard I, Cassier P, Decouvelaere AV, Ranchere D, Kurtz JE, Bergerat JP, Blay JY. Insulin-like growth factor type 1 receptor (IGF-1R) exclusive nuclear staining: a predictive biomarker for IGF-1R monoclonal antibody (Ab) therapy in sarcomas. Eur J Cancer. 2012 Nov;48(16):3027-35. doi: 10.1016/j.ejca.2012.05.009. Epub 2012 Jun 7. PMID 22682017
- [Derived] Pappo AS, Patel SR, Crowley J, Reinke DK, Kuenkele KP, Chawla SP, Toner GC, Maki RG, Meyers PA, Chugh R, Ganjoo KN, Schuetze SM, Juergens H, Leahy MG, Geoerger B, Benjamin RS, Helman LJ, Baker LH. R1507, a monoclonal antibody to the insulin-like growth factor 1 receptor, in patients with recurrent or refractory Ewing sarcoma family of tumors: results of a phase II Sarcoma Alliance for Research through Collaboration study. J Clin Oncol. 2011 Dec 1;29(34):4541-7. doi: 10.1200/JCO.2010.34.0000. Epub 2011 Oct 24. PMID 22025149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A screening period was included prior to administration of study drug. Tumor scans/X-rays were to be obtained within 4 weeks, fluro-D-glucose positron emission tomography (FDG-PET) scans within 2 weeks, and Baseline laboratory evaluations within 1 week before first dose.
Groups:
- Cohort 7a: Alveolar Soft Part Sarcoma: Participants 2 years of age and older with recurrent or refractory sarcoma received R1507 as 9 mg/kg via IV infusion once weekly until disease progression, intercurrent illness, unacceptable toxicity, prolonged (2-week) time off treatment, withdrawal, loss to follow-up, investigator decision, or death. Cohort 7a included individuals with alveolar soft part sarcoma.
Period: Overall Study
Arm/Group | Cohort 1: Ewings Sarcoma Primary Cohort | Cohort 2: Ewings Sarcoma Secondary Cohort | Cohort 3: Ewings Sarcoma Expanded Cohort | Cohort 4: Osteosarcoma | Cohort 5: Synovial Sarcoma | Cohort 6: Rhabdomyosarcoma | Cohort 7a: Alveolar Soft Part Sarcoma | Cohort 7b: Desmoplastic Small Round Cell Tumors. | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma | Cohort 7d: Clear Cell Sarcoma | Cohort 7e: Myxoid Liposarcoma | Cohort 8: Diagnosis Not Specified
Started | 70 | 54 | 7 | 40 | 25 | 41 | 23 | 14 | 11 | 9 | 12 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 70 | 54 | 7 | 40 | 25 | 41 | 23 | 14 | 11 | 9 | 12 | 11
Not completed — Physician Decision | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Death | 4 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study closed by Sponsor | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Other | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Disease progression | 60 | 50 | 5 | 36 | 23 | 39 | 18 | 12 | 10 | 7 | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Ewings Sarcoma Primary Cohort | Cohort 2: Ewings Sarcoma Secondary Cohort | Cohort 3: Ewings Sarcoma Expanded Cohort | Cohort 4: Osteosarcoma | Cohort 5: Synovial Sarcoma | Cohort 6: Rhabdomyosarcoma | Cohort 7a: Alveolar Soft Part Sarcoma | Cohort 7b: Desmoplastic Small Round Cell Tumors. | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma | Cohort 7d: Clear Cell Sarcoma | Cohort 7e: Myxoid Liposarcoma | Cohort 8: Diagnosis Not Specified | Total
Number analyzed (Participants) | 70 | 54 | 7 | 40 | 25 | 41 | 23 | 14 | 11 | 9 | 12 | 11 | 317
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27 (10.72) | 28.3 (12.9) | 13.3 (3.15) | 33.8 (18.83) | 41.7 (16.11) | 26.5 (12.21) | 31.7 (13.67) | 23.1 (6.09) | 60.9 (11.27) | 26.9 (11.01) | 50.6 (11.06) | 30.7 (18.56) | 31.2 (13.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 3 | 20 | 11 | 18 | 12 | 1 | 3 | 2 | 3 | 3 | 118
  Male | 50 | 32 | 4 | 20 | 14 | 23 | 11 | 13 | 8 | 7 | 9 | 8 | 199

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete or Partial Response, According to World Health Organization (WHO) Criteria in Cohorts 2 to 8
Description: Complete response is the disappearance of all known disease, determined by two consecutive observations not less than 4 weeks apart. Partial response is >=50% decrease in the total tumor load of the lesions that have been measured to determine the effect of therapy not less than four weeks apart. The observations must be consecutive.
Time Frame: Baseline up to 6 years (assessed at baseline, every 6 weeks for 24 weeks, then every 12 weeks until disease progression)
Population: ITT population included all randomized participants who received at least 1 dose of study drug and had at least 1 post baseline efficacy assessment. There were 0 participants analyzed for Cohort 3 due to no efficacy data being collected for that cohort.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 2: Ewings Sarcoma Secondary Cohort | Cohort 3: Ewings Sarcoma Expanded Cohort | Cohort 4: Osteosarcoma | Cohort 5: Synovial Sarcoma | Cohort 6: Rhabdomyosarcoma | Cohort 7a: Alveolar Soft Part Sarcoma | Cohort 7b: Desmoplastic Small Round Cell Tumors. | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma | Cohort 7d: Clear Cell Sarcoma | Cohort 7e: Myxoid Liposarcoma | Cohort 8: Diagnosis Not Specified
Number analyzed (Participants) | 54 | 0 | 40 | 25 | 41 | 23 | 14 | 11 | 9 | 12 | 11
Percentage of Participants | 11.11 |  | 2.5 | 4.0 | 4.88 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Progression-Free Survival (PFS) Rate According to WHO Response Criteria at 18 Weeks From Start of R2607 Treatment in Cohort 1
Description: The PFS survival rate is a landmark analysis of progression-free survival at 18 weeks from start of treatment. Progression-free survival rate at 18 weeks is a dichotomous endpoint, with a patient categorized as alive (with either stable disease or objective response) at 18 weeks from start of treatment.
Time Frame: Baseline up to 18 weeks (assessed at baseline, every 6 weeks until disease progression)
Population: ITT population included all randomized participants who received at least 1 dose of study drug and had at least 1 post baseline efficacy assessment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: Ewings Sarcoma Primary Cohort
Number analyzed (Participants) | 70
Percentage of Participants | 15.81

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs) in Cohort 1 and 2
Time Frame: Baseline up to 6 years
Population: Safety Population: All participants who received at least one dose of study drug at had at least one safety follow-up assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Ewings Sarcoma Primary Cohort | Cohort 2: Ewings Sarcoma Secondary Cohort
Number analyzed (Participants) | 70 | 54
percentage of participants | 96 | 96

4. Secondary Outcome: Percentage of Participants With Complete or Partial Response According to WHO Response Criteria in Cohort 1
Description: as for outcome 1
Time Frame: Baseline, every 6 weeks for 24 weeks, then every 12 weeks until disease progression (up to 6 years)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Ewings Sarcoma Primary Cohort
Number analyzed (Participants) | 70
percentage of participants | 8.57

5. Secondary Outcome: PFS Rate According to WHO Response Criteria at 18 Weeks From Start of R1507 Treatment in Cohorts 2 to 8
Description: The PFS survival rate is a landmark analysis of progression-free survival at 18 weeks from start of treatment. Progression-free survival rate at 18 weeks is a dichotomous endpoint, with a patient categorized as alive (with either stable disease or objective response at 18 weeks) from start of treatment.
Time Frame: Baseline, every 6 weeks until disease progression (up to 18 weeks)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 2: Ewings Sarcoma Secondary Cohort | Cohort 3: Ewings Sarcoma Expanded Cohort | Cohort 4: Osteosarcoma | Cohort 5: Synovial Sarcoma | Cohort 6: Rhabdomyosarcoma | Cohort 7a: Alveolar Soft Part Sarcoma | Cohort 7b: Desmoplastic Small Round Cell Tumors. | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma | Cohort 7e: Myxoid Liposarcoma | Cohort 7d: Clear Cell Sarcoma | Cohort 8: Diagnosis Not Specified
Number analyzed (Participants) | 54 | 0 | 40 | 25 | 41 | 23 | 14 | 11 | 9 | 12 | 11
Percentage of Participants | 17.16 |  | 19.69 | 4.00 | 7.32 | 45.40 | 8.16 | 62.34 | 0 | 8.33 | 22.86

6. Secondary Outcome: Percentage of Participants With AEs in Cohorts 3-8
Time Frame: Baseline up to 6 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 3: Ewings Sarcoma Expanded Cohort | Cohort 4: Osteosarcoma | Cohort 5: Synovial Sarcoma | Cohort 6: Rhabdomyosarcoma | Cohort 7a: Alveolar Soft Part Sarcoma | Cohort 7b: Desmoplastic Small Round Cell Tumors. | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma | Cohort 7d: Clear Cell Sarcoma | Cohort 7e: Myxoid Liposarcoma | Cohort 8: Diagnosis Not Specified
Number analyzed (Participants) | 7 | 40 | 25 | 41 | 23 | 14 | 11 | 9 | 12 | 11
percentage of participants | 85.7 | 100 | 100 | 95 | 91 | 86 | 100 | 100 | 100 | 100

7. Secondary Outcome: Duration of Response (DOR) According to WHO Response Criteria in Cohorts 1 to 8
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Complete response is the disappearance of all known disease, determined by two consecutive observations not less than 4 weeks apart. Partial response is >=50% decrease in the total tumor load of the lesions that have been measured to determine the effect of therapy not less than four weeks apart. The observations must be consecutive.
Time Frame: Baseline, every 6 weeks for 24 weeks, then every 12 weeks until disease progression (up to 6 years)
Population: ITT population included all randomized participants who received at least 1 dose of study drug and had at least 1 post baseline efficacy assessment. There were 0 participants analyzed for Cohort 3, 7 and 8 due to no DOR data being collected for these cohorts.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1: Ewings Sarcoma Primary Cohort | Cohort 2: Ewings Sarcoma Secondary Cohort | Cohort 3: Ewings Sarcoma Expanded Cohort | Cohort 4: Osteosarcoma | Cohort 5: Synovial Sarcoma | Cohort 6: Rhabdomyosarcoma | Cohort 7a: Alveolar Soft Part Sarcoma | Cohort 7b: Desmoplastic Small Round Cell Tumors. | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma | Cohort 7d: Clear Cell Sarcoma | Cohort 7e: Myxoid Liposarcoma | Cohort 8: Diagnosis Not Specified
Number analyzed (Participants) | 70 | 54 | 0 | 40 | 25 | 41 | 0 | 0 | 0 | 0 | 0 | 0
weeks | 44.29 [18 to NA] — Upper limit was not reached due to low number of events. | 42.86 [18.14 to NA] — Upper limit was not reached due to low number of events. |  | NA [30.14 to NA] — DOR and upper limit were not reached due to low number of events. | 13.14 [13.14 to NA] — Upper limit was not reached due to low number of events. | NA [21 to NA] — DOR and upper limit were not reached due to low number of events. |  |  |  |  |  |

8. Secondary Outcome: Time to Progression (TTP) According to WHO Response Criteria in Cohorts 1 to 8
Description: TTP is defined as the time from date of randomization until objective tumor progression. According to the WHO Response Criteria, objective tumor progression is > 25% increase in the area of one or more measurable lesions or the appearance of new lesions.
Time Frame: Baseline, every 6 weeks for 24 weeks, then every 12 weeks until disease progression (up to 6 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1: Ewings Sarcoma Primary Cohort | Cohort 2: Ewings Sarcoma Secondary Cohort | Cohort 3: Ewings Sarcoma Expanded Cohort | Cohort 4: Osteosarcoma | Cohort 5: Synovial Sarcoma | Cohort 6: Rhabdomyosarcoma | Cohort 7a: Alveolar Soft Part Sarcoma | Cohort 7b: Desmoplastic Small Round Cell Tumors. | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma | Cohort 7d: Clear Cell Sarcoma | Cohort 7e: Myxoid Liposarcoma | Cohort 8: Diagnosis Not Specified
Number analyzed (Participants) | 70 | 54 | 0 | 40 | 25 | 41 | 23 | 14 | 11 | 9 | 12 | 11
weeks | 6.00 [5.29 to 9.71] | 6.00 [5.71 to 8.14] |  | 5.71 [5.57 to 7.00] | 6.00 [5.57 to 6.43] | 5.50 [5.14 to 6.14] | 11.14 [6.00 to 17.71] | 6.14 [5.86 to 11.14] | 18.00 [5.71 to NA] — Upper limit was not reached due to low number of events. | 5.57 [5.14 to 5.86] | 5.86 [5.29 to 8.43] | 6.14 [5.86 to 10.00]

9. Secondary Outcome: Failure-Free Survival (FFS) According to WHO Response Criteria in Cohorts 1 to 8
Description: FFS was measured from the date of treatment start to the date of documented disease progression, relapse, or death from any cause.
Time Frame: Baseline, every 6 weeks for 24 weeks, then every 12 weeks until disease progression (up to 6 years)
Population: Data was not collected for this endpoint.
Arm/Group | Cohort 1: Ewings Sarcoma Primary Cohort | Cohort 2: Ewings Sarcoma Secondary Cohort | Cohort 3: Ewings Sarcoma Expanded Cohort | Cohort 4: Osteosarcoma | Cohort 5: Synovial Sarcoma | Cohort 6: Rhabdomyosarcoma | Cohort 7a: Alveolar Soft Part Sarcoma | Cohort 7b: Desmoplastic Small Round Cell Tumors. | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma | Cohort 7d: Clear Cell Sarcoma | Cohort 7e: Myxoid Liposarcoma | Cohort 8: Diagnosis Not Specified
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Overall Survival (OS) in Cohorts 1 to 8
Description: OS was measured from the time of study registration to the date of death or was censored at the date of last contact.
Time Frame: Baseline until death (up to 6 years)
Population: ITT population included all randomized participants who received at least 1 dose of study drug and had at least 1 post baseline efficacy assessment. There were 0 participants analyzed for Cohort 3 and 7c due to no overall survival data being collected for those cohorts.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1: Ewings Sarcoma Primary Cohort | Cohort 2: Ewings Sarcoma Secondary Cohort | Cohort 3: Ewings Sarcoma Expanded Cohort | Cohort 4: Osteosarcoma | Cohort 5: Synovial Sarcoma | Cohort 6: Rhabdomyosarcoma | Cohort 7a: Alveolar Soft Part Sarcoma | Cohort 7b: Desmoplastic Small Round Cell Tumors. | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma | Cohort 7d: Clear Cell Sarcoma | Cohort 7e: Myxoid Liposarcoma | Cohort 8: Diagnosis Not Specified
Number analyzed (Participants) | 70 | 54 | 0 | 40 | 25 | 61 | 23 | 14 | 11 | 9 | 12 | 11
weeks | 29.57 [20.57 to 37.57] | 43.57 [33.29 to 69.00] |  | 37.14 [25.57 to NA] — Upper limit was not reached due to low number of events. | 40.71 [21.71 to 64.14] | 30.86 [21.57 to 50.00] | 42.43 [42.43 to NA] — Upper limit was not reached due to low number of events. | 40.86 [23.57 to NA] — Upper limit was not reached due to low number of events. | NA [NA to NA] — All participants were censored as no deaths occurred. | 17.00 [9.14 to NA] — Upper limit was not reached due to low number of events. | 36.00 [33.14 to NA] — Upper limit was not reached due to low number of events. | 17.43 [13.00 to 30.14]

11. Secondary Outcome: PFS According to WHO Response Criteria in Cohorts 1 to 8
Description: PFS is defined as the duration of time from start of treatment to time of objective progression or death.
Time Frame: Baseline, every 6 weeks for 24 weeks, then every 12 weeks until disease progression (up to 6 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1: Ewings Sarcoma Primary Cohort | Cohort 2: Ewings Sarcoma Secondary Cohort | Cohort 3: Ewings Sarcoma Expanded Cohort | Cohort 4: Osteosarcoma | Cohort 5: Synovial Sarcoma | Cohort 6: Rhabdomyosarcoma | Cohort 7a: Alveolar Soft Part Sarcoma | Cohort 7b: Desmoplastic Small Round Cell Tumors. | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma | Cohort 7d: Clear Cell Sarcoma | Cohort 7e: Myxoid Liposarcoma | Cohort 8: Diagnosis Not Specified
Number analyzed (Participants) | 70 | 54 | 0 | 40 | 25 | 41 | 23 | 14 | 11 | 9 | 12 | 11
weeks | 6.00 [5.29 to 9.57] | 6.00 [5.71 to 8.14] |  | 5.71 [5.57 to 6.43] | 6.00 [5.43 to 6.14] | 5.43 [5.14 to 6.14] | 11.14 [5.71 to 11.71] | 6.14 [5.86 to 11.14] | 18.00 [5.71 to NA] — Upper limit was not reached due to low number of events. | 5.57 [5.14 to 5.86] | 5.86 [5.29 to 8.43] | 6.14 [5.86 to 10]

12. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) of R1507
Time Frame: Predose (0 hours [h]), end of 60-90 minutes infusion (EOI), postdose (2, 24, 72-96 h) in Week 1; predose (0 h) and EOI in Weeks 2, 4, 6, 9; predose (0 h), EOI, postdose (48 h) in Week 12; predose (0 h) in Week 13, at final visit (up to 6 years)
Population: Data was not collected for this pharmacokinetic endpoint.
Arm/Group | Cohort 1: Ewings Sarcoma Primary Cohort | Cohort 2: Ewings Sarcoma Secondary Cohort | Cohort 3: Ewings Sarcoma Expanded Cohort | Cohort 4: Osteosarcoma | Cohort 5: Synovial Sarcoma | Cohort 6: Rhabdomyosarcoma | Cohort 7a: Alveolar Soft Part Sarcoma | Cohort 7b: Desmoplastic Small Round Cell Tumors. | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma | Cohort 7d: Clear Cell Sarcoma | Cohort 7e: Myxoid Liposarcoma | Cohort 8: Diagnosis Not Specified
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Pharmacokinetics: Clearance (CL) of R1507
Time Frame: Predose (0 h), EOI (infusion over 60-90 minutes), postdose (2, 24, 72-96 h) in Week 1; predose (0 h) and EOI in Weeks 2, 4, 6, 9; predose (0 h), EOI, postdose (48 h) in Week 12; predose (0 h) in Week 13, at final visit (up to 6 years)
Population: Data was not collected for this pharmacokinetic endpoint.
Arm/Group | Cohort 1: Ewings Sarcoma Primary Cohort | Cohort 2: Ewings Sarcoma Secondary Cohort | Cohort 3: Ewings Sarcoma Expanded Cohort | Cohort 4: Osteosarcoma | Cohort 5: Synovial Sarcoma | Cohort 6: Rhabdomyosarcoma | Cohort 7a: Alveolar Soft Part Sarcoma | Cohort 7b: Desmoplastic Small Round Cell Tumors. | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma | Cohort 7d: Clear Cell Sarcoma | Cohort 7e: Myxoid Liposarcoma | Cohort 8: Diagnosis Not Specified
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 6 years
Description: Safety Population: All participants who received at least one dose of study drug at had at least one safety follow-up assessment.
Arm/Group | Cohort 1: Ewings Sarcoma Primary Cohort | Cohort 2: Ewings Sarcoma Secondary Cohort | Cohort 3: Ewings Sarcoma Expanded Cohort | Cohort 4: Osteosarcoma | Cohort 5: Synovial Sarcoma | Cohort 6: Rhabdomyosarcoma | Cohort 7a: Alveolar Soft Part Sarcoma | Cohort 7b: Desmoplastic Small Round Cell Tumors | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma | Cohort 7d: Clear Cell Sarcoma | Cohort 7e: Myxoid Liposarcoma | Cohort 8: Diagnosis Not Specified
All-Cause Mortality (participants affected / at risk) | 9/70 | 5/54 | 2/7 | 7/40 | 3/25 | 3/41 | 1/23 | 0/14 | 0/11 | 1/9 | 1/12 | 2/11
Serious Adverse Events (participants affected / at risk) | 11/70 | 13/54 | 1/7 | 4/40 | 5/25 | 4/41 | 1/23 | 1/14 | 0/11 | 3/9 | 2/12 | 4/11
Other Adverse Events (participants affected / at risk) | 67/70 | 52/54 | 6/7 | 40/40 | 25/25 | 39/41 | 21/23 | 12/14 | 11/11 | 9/9 | 12/12 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ewings Sarcoma Primary Cohort (N=70) | Cohort 2: Ewings Sarcoma Secondary Cohort (N=54) | Cohort 3: Ewings Sarcoma Expanded Cohort (N=7) | Cohort 4: Osteosarcoma (N=40) | Cohort 5: Synovial Sarcoma (N=25) | Cohort 6: Rhabdomyosarcoma (N=41) | Cohort 7a: Alveolar Soft Part Sarcoma (N=23) | Cohort 7b: Desmoplastic Small Round Cell Tumors (N=14) | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma (N=11) | Cohort 7d: Clear Cell Sarcoma (N=9) | Cohort 7e: Myxoid Liposarcoma (N=12) | Cohort 8: Diagnosis Not Specified (N=11)
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adrenal haemorrhage (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ewings Sarcoma Primary Cohort (N=70) | Cohort 2: Ewings Sarcoma Secondary Cohort (N=54) | Cohort 3: Ewings Sarcoma Expanded Cohort (N=7) | Cohort 4: Osteosarcoma (N=40) | Cohort 5: Synovial Sarcoma (N=25) | Cohort 6: Rhabdomyosarcoma (N=41) | Cohort 7a: Alveolar Soft Part Sarcoma (N=23) | Cohort 7b: Desmoplastic Small Round Cell Tumors (N=14) | Cohort 7c: Extraskeletal Myxoid Chondrosarcoma (N=11) | Cohort 7d: Clear Cell Sarcoma (N=9) | Cohort 7e: Myxoid Liposarcoma (N=12) | Cohort 8: Diagnosis Not Specified (N=11)
Alanine aminotransferase increased (Investigations) | 5 | 2 | 1 | 2 | 3 | 7 | 2 | 2 | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 4 | 1 | 5 | 4 | 5 | 1 | 1 | 0 | 0 | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 8 | 2 | 0 | 5 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 5 | 2 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 1 | 1 | 2
Weight decreased (Investigations) | 8 | 6 | 0 | 6 | 1 | 4 | 4 | 1 | 2 | 2 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 0 | 9 | 5 | 3 | 6 | 0 | 6 | 3 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 13 | 0 | 5 | 4 | 2 | 1 | 1 | 1 | 2 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0 | 3 | 0 | 3 | 4 | 1 | 2 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 0 | 5 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 8 | 5 | 0 | 4 | 1 | 3 | 2 | 1 | 0 | 2 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 4 | 0 | 3 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 10 | 17 | 0 | 4 | 0 | 7 | 5 | 3 | 1 | 1 | 1 | 4
Asthenia (General disorders) | 5 | 9 | 0 | 4 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 4
Chest pain (General disorders) | 7 | 7 | 0 | 6 | 3 | 2 | 3 | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 19 | 22 | 1 | 13 | 3 | 14 | 5 | 5 | 5 | 5 | 5 | 3
Infusion related reaction (General disorders) | 5 | 3 | 0 | 4 | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 11 | 6 | 1 | 1 | 0 | 4 | 1 | 2 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 10 | 13 | 0 | 3 | 3 | 0 | 6 | 2 | 0 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 4 | 1 | 0 | 5 | 3 | 4 | 0 | 3 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 0 | 2 | 2 | 4 | 1 | 3 | 0 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 12 | 10 | 0 | 7 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 15 | 0 | 8 | 3 | 6 | 7 | 1 | 3 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 9 | 20 | 0 | 7 | 5 | 10 | 6 | 1 | 2 | 4 | 3 | 3
Vomiting (Gastrointestinal disorders) | 11 | 11 | 0 | 8 | 4 | 8 | 6 | 0 | 1 | 2 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 6 | 0 | 1 | 1 | 3 | 1 | 2 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6 | 0 | 2 | 0 | 2 | 2 | 0 | 2 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 8 | 0 | 9 | 1 | 6 | 4 | 3 | 2 | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 0 | 5 | 1 | 0 | 1 | 1 | 1 | 3 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 13 | 12 | 0 | 2 | 1 | 7 | 2 | 2 | 3 | 2 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 9 | 0 | 5 | 4 | 4 | 4 | 3 | 5 | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 3 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2 | 1 | 1 | 2 | 1 | 4 | 0 | 0 | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 7 | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 3 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 4 | 3 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 4 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 1 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 0
Haemoglobin (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Aspartate Aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Blood alkaline phosphatase (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood creatinine (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
White blood cell count (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematocrit (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urine bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 2 | 2 | 3 | 2 | 0 | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 4 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 6 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Borrelia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 5 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Haemoglobinaemia (Blood and lymphatic system disorders) | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 4 | 0 | 1 | 0 | 3 | 2 | 1 | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 5 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Decreased activity (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 3 | 0 | 2 | 0
Hot flush (Vascular disorders) | 1 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pericardia effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 3 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 4 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 0 | 3 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 3 | 1 | 0 | 3 | 3 | 0 | 2 | 0 | 0 | 0 | 3 | 2
Oedema (General disorders) | 4 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Chills (General disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyperthermia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was closed to further enrollment due to a decision by the Sponsor to discontinue development of R1507. The decision was made based upon available data from other completed/ongoing trials of R1507 and was not due to safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.